CLINICAL TRIAL: NCT04302467
Title: Effects of Goal-directed Fluid Therapy and Restrictive Fluid Therapy During Operation Combined With Enhanced Recovery After Surgery Protocol on Acute Kidney Injury After Thoracoscopic Lobectomy in High Risk Patients
Brief Title: Effects of Intraoperative Fluid Therapy on Acute Kidney Injury After Thoracoscopic Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJTU1AF-CRF-2019-012
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2021-08

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Goal-directed fluid therapy; Enhanced recovery after surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of the two groups: (1) GDFT group and (2) restrictive fluid therapy group. They will be allocated in a 1:1 ratio using random numbers generated by Microsoft Excel.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocations will be blinded to all participants but the anesthesiologists. If serious adverse events occur, the patients will be removed from the trial, the blinding will be removed, the events will be reported to the institutional review board.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDFT group (Experimental): Fluid maintenance with 2 ml/kg/h of Ringer's solution of sodium acetate, when SVV>13%, 4 mL/kg bolus of hydroxyethyl starch will be infused within 5 min. If SVV falls below 13%, the bolus will be suspended. If SVV is still more than 13%, 100 μg of phenylephrine will be administered when CI is more than 2.5 L/min/m2, 1 mg of dopamine will be administered when CI is less than 2.5 L/min/m2. When SVV<13%, but mean arterial pressure (MAP)<65 mmHg, 8 μg of norepinephrine will be administered. The hemodynamic status will be repeatedly measured every 10 min.
  Interventions: Procedure: fluid therapy during operation
- restrictive fluid therapy group (Experimental): fluid maintenance with 2 ml/kg/h of Ringer's solution of sodium acetate, hydroxyethyl starch will be infused to supply blood loss, the ratio of hydroxyethyl starch to blood loss is 1:1. 0.01-0.1 μg/kg/min of norepinephrine will be administered to maintain MAP>65 mmHg.
  Interventions: Procedure: fluid therapy during operation

INTERVENTIONS:
Procedure: fluid therapy during operation — ERAS protocol of lobectomy will implemented to all the participants during perioperation,two groups of participants will be given different intraoperative fluid therapy strategy.
  Other Names: Implement ERAS protocol of lobectomy during perioperation

SUMMARY:
Background: Acute kidney injury (AKI) often occurs after thoracoscopic lobectomy in high risk patients. Insufficient intraoperative infusion is risk factor of AKI. Goal-directed fluid therapy (GDFT) is individualized fluid infusion strategy, the infusion rate and type is adjusted according to the individual's fluid response. GDFT during operation can reduce the incidence of AKI after major surgery. Enhanced recovery after surgery (ERAS) integrates a range of perioperative interventions to decrease postoperative complications after surgery. In ERAS protocol of lobectomy, restrictive fluid therapy during operation is recommended. In this study, the investigators will compare the effects of GDFT and restrictive fluid therapy during operation combined with ERAS protocol on the incidence of AKI after thoracoscopic lobectomy in high risk patients.

Methods/design: This is prospective single-center single-blind randomized controlled trial. 276 patients scheduled to undergo thoracoscopic lobectomy under general anesthesia combined with paravertebral block are randomly divided into GDFT group and restrictive fluid therapy group at a 1:1 ratio. The primary outcome is the incidence of AKI after operation. The secondary outcomes are (1) the incidence of renal replacement therapy, (2) length of intensive care unit (ICU) stay after operation, (3) length of hospital stay after operation , (4) incidence of other complications including: infection, acute lung injury (ALI), pneumonia, arrhythmia, heart failure, myocardial injury after noncardiac surgery (MINS), cardiac infarction.

Discussion: This is the first study to compare GDFT and restrictive fluid therapy during operation combined with ERAS protocol on the incidence of AKI after thoracoscopic lobectomy in high risk patients. The investigators expected that the two methods have the same effect on the incidence of AKI, but restrictive fluid therapy is simpler to applied than GDFT.

DETAILED DESCRIPTION:
Participants: Patients aged more than 18 years old who are scheduled to undergo thoracoscopic lobectomy well be enrolled in this trial. Participants will be randomly allocated to one of the two groups: (1) GDFT group and (2) restrictive fluid therapy group. Participants will be allocated in a 1:1 ratio using random numbers generated by Microsoft Excel.

Interventions: All participants will start lung function exercise, quit smoking, reinforce nutrition after hospitalization. Participants will fast for 6 hours and prohibit of drinking water for 2 hours before operation. Antibiotic will be used 1 hour before operation. No premedication will be administered to the patients. The electrocardiography (ECG), pulse oximetry, invasive arterial blood pressure, nasopharyngeal temperature, and bispectral index monitoring will be instituted. Urinary catheter will be inserted after anesthesia and removed immediately after operation. Patients will undergo thoracoscopic lobectomy under general anesthesia combined with paravertebral block. General anesthesia will be inducted with sufentanil, propofol, and rocuronium, and maintained with continuous infusion of propofol and remifentanil, intermittent injection of rocuronium. Lung-protective ventilation strategy will be used during mechanical ventilation. Recovery from general anesthesia as quickly as possible. Paravertebral block will be performed under the guidance of ultrasound after general anesthesia induction. Paravertebral block, patient controlled analgesia and oral analgesics will be used for postoperative analgesia. Recovering of oral rehydration, eating and getting out of bed as early as possible.

In GDFT group, the arterial catheter will be connected with FloTrac/Vigileo sensor (Edwards lifesciences, Irvine, CA, USA), The stroke volume variation (SVV) and cardiac index (CI) will be monitored. Fluid maintenance with 2 ml/kg/h of Ringer's solution of sodium acetate, when SVV>13%, 4 mL/kg bolus of hydroxyethyl starch will be infused within 5 min. If SVV falls below 13%, the bolus will be suspended. If SVV is still more than 13%, 100 μg of phenylephrine will be administered when CI is more than 2.5 L/min/m2, 1 mg of dopamine will be administered when CI is less than 2.5 L/min/m2. When SVV<13%, but mean arterial pressure (MAP)<65 mmHg, 8 μg of norepinephrine will be administered. The hemodynamic status will be repeatedly measured every 10 min.

In restrictive fluid therapy group, fluid maintenance with 2 ml/kg/h of Ringer's solution of sodium acetate, hydroxyethyl starch will be infused to supply blood loss, the ratio of hydroxyethyl starch to blood loss is 1:1. 0.01-0.1 μg/kg/min of norepinephrine will be administered to maintain MAP>65 mmHg.

Measurements: The primary outcome is the incidence of AKI after operation. The secondary outcomes include: (1) Incidence of renal replacement therapy, (2) Length of ICU stay after operation, (3) Length of hospital stay after operation, (4) Incidence of other complications including: infection, ALI, pneumonia, arrhythmia, heart failure, MINS, cardiac infarction.

Sample size: The primary outcome of this trial is the incidence of AKI after operation. Another study showed that the incidence of AKI was 4% and 2.9% in liberal infusion and GDFT respectively, the efficacy of intervention was 27.5%. Investigators hypothesis that restrictive fluid therapy combined with ERAS protocol has the same therapeutic effect as GDFT. The sample size for this study was calculated to achieve a statistical power of 0.8 and alpha error of 0.05 using a two-sided test. Considering a dropout rate of 10%, 138 patients are required in each group.

Statistical analysis: Normally distributed data will be presented as the mean±standard deviation. Categorical data will be presented as the number and the percentage of patients. The primary outcome (the incidence of AKI after operation) will be compared between the two groups with Pearson's chi-square test. The secondary outcomes will be compared between the two groups with independent-samples Student's t-tests for normally distributed continuous data and Pearson's chi-square test for categorical data. All statistical test are two-sided, and a P-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: patients comply any of the following criteria will be enrolled

* Age>70 years old
* Forced expiratory volume in 1 second (FEV1)<60%
* Carbon monoxide lung diffusion capacity (DLCO)<60%
* History of coronary artery disease

Exclusion Criteria: patients comply any of the following criteria may not be enrolled

* Patients refused
* Creatinine>176 μmol/L, and/or BUN>7.1 mmol/L
* NT-proBNP>300 ng/L
* Systemic or local infection
* Albumin<30 g/L, and/or Hemoglobin<100 g/L
* Allergy to hydroxyethyl starch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
number of participants with acute kidney injury | 48 hours after operation
  50% relative or 0.3 mg/dl (26.5 μmol/L) absolute increase in creatinine over the preoperative value during the first two postoperative days.

SECONDARY OUTCOMES:
number of participants in need of renal replacement therapy | 30 days after operation
  Patients who need renal replacement therapy, the indications of renal replacement therapy will be determined by clinician
length of ICU stay after operation | 30 days after operation
  from the end of operation to ICU discharge
length of hospital stay after operation | 30 days after operation
  from the end of operation to discharge
number of participants with infection | 30 days after operation
  Patients with postoperative infection, including: wound infection, urinary tract infection, systemic infection
number of participants with acute lung injury | 24 hours after operation
  Oxygen partial pressure/fraction of inhaled oxygen(PaO2/FiO2)<300 mmHg 24 hours after operation, bilateral lung infiltration, exclude cardiogenic pulmonary edema.
number of participants with pneumonia | 30 days after operation
  new or progressive and persistent infiltrates, consolidation, cavitation. And at least one of the following: (1) fever (>38℃) with no other recognised cause, (2) white cell count<4×109/L or >12×109/L, (3) altered mental status with no other recognised cause for patients more than 70 years old. And at least two of the following:(1) new onset of purulent sputum or change in character of sputum, or increased respiratory secretions, or increased suctioning requirements, (2) new onset or worsening cough, or dyspnea, or tachypnea, (3) rales or bronchial breath sounds, (4) worse gas exchange.
number of participants with arrhythmia | 48 hours after operation
  patients who have new-onset arrhythmia 48 hours after operation
number of participants with heart failure | 48 hours after operation
  NT-proBNP is more than 450 ng/L if age less than 50, or NT-proBNP is more than 900 ng/L if age more than 50.
number of participants with myocardial injury after noncardiac surgery | 7 days after operation
  troponin T is more than 0.03 ng/ml and/or creatine kinase-MB is more than 8.8 ng/ml.
number of participants with cardiac infarction | 48 hours after operation
  troponin T elevation in the presence of at least one of ischemic symptoms: (1) the development of new or presumed new Q waves, (2) ST segment or T wave changes, (3) left bundle branch block on ECG, (4) a new or presumed new regional wall motion abnormality on echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Guan, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Participants' private information will not be collected. Only the study code will be collected. The data collected will be kept confidential until they are required for analysis. The data collected will be stored under encryption for 2 years after the completion of the study.

REFERENCES:
- [Derived] Ma H, Li X, Wang Z, Qiao Q, Gao Y, Yuan H, Guan B, Guan Z. The effect of intraoperative goal-directed fluid therapy combined with enhanced recovery after surgery program on postoperative complications in elderly patients undergoing thoracoscopic pulmonary resection: a prospective randomized controlled study. Perioper Med (Lond). 2023 Jul 10;12(1):33. doi: 10.1186/s13741-023-00327-x. PMID 37430359
- [Derived] Guan Z, Gao Y, Qiao Q, Wang Q, Liu J. Effects of intraoperative goal-directed fluid therapy and restrictive fluid therapy combined with enhanced recovery after surgery protocol on complications after thoracoscopic lobectomy in high-risk patients: study protocol for a prospective randomized controlled trial. Trials. 2021 Jan 7;22(1):36. doi: 10.1186/s13063-020-04983-y. PMID 33413593